CLINICAL TRIAL: NCT00104910
Title: A Phase I Trial of Tailored Radiation Therapy With Concomitant Cetuximab (C225, NSC #714692) and Cisplatin (NSC #119875) in the Treatment of Patients With Cervical Cancer
Brief Title: Cetuximab, Cisplatin, and Radiation Therapy in Treating Patients With Stage IB, Stage II, Stage III, or Stage IVA Cervical Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: GOG Foundation (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GOG-9918; NCI-2009-00621 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000413880; GOG-9918; GOG-9918 (Other: Gynecologic Oncology Group); GOG-9918 (Other: CTEP); U10CA027469 (NIH)
Record Dates: First submitted 2005-03-03; First posted 2005-03-04 (Estimated); Last update posted 2014-12-31 (Estimated); Status verified 2014-12

CONDITIONS: Cervical Adenocarcinoma; Cervical Adenosquamous Carcinoma; Cervical Small Cell Carcinoma; Cervical Squamous Cell Carcinoma; Stage IB Cervical Cancer; Stage IIA Cervical Cancer; Stage IIB Cervical Cancer; Stage III Cervical Cancer; Stage IVA Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Brachytherapy; Radiotherapy, Conformal; Cetuximab; Cisplatin

ARMS (1):
- Treatment (brachytherapy, radiation, cetuximab, cisplatin) (Experimental): Patients receive cetuximab IV over 1-2 hours and cisplatin IV on days 1, 8, 15, 22, 29, and 36 (weeks 1-6). Patients also undergo external beam radiotherapy to the para-aortic and pelvic lymph nodes OR whole pelvis once daily on days 1-5, 8-12, 15-19, 22-26, and 29-33 (weeks 1-5). Patients then receive either 1 or 2 applications of low-dose rate brachytherapy in weeks 6-8 OR 5 applications of high-dose rate (HDR)* brachytherapy once weekly in weeks 4-8. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Radiation: Internal Radiation Therapy; Radiation: 3-Dimensional Conformal Radiation Therapy; Biological: Cetuximab; Drug: Cisplatin

INTERVENTIONS:
Radiation: Internal Radiation Therapy
  Other Names: Brachytherapy; Internal Radiation; Internal Radiation Brachytherapy; Radiation Brachytherapy
Radiation: 3-Dimensional Conformal Radiation Therapy
  Other Names: 3D-CRT; Conformal Therapy; Radiation Conformal Therapy
Biological: Cetuximab — Given IV
  Other Names: Chimeric MoAb C225; Erbitux; IMC-C225
Drug: Cisplatin — Given IV

SUMMARY:
This phase I trial is studying the side effects and best dose of cetuximab when given together with cisplatin and radiation therapy in treating patients with stage IB, stage II, stage III, or stage IVA cervical cancer. Monoclonal antibodies, such as cetuximab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Drugs used in chemotherapy, such as cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays and other types of radiation to kill tumor cells. Internal radiation therapy uses radioactive material placed directly into or near a tumor to kill tumor cells. Giving cetuximab together with cisplatin and radiation therapy may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the maximum tolerated dose or safe biologically effective dose of cetuximab when administered in combination with cisplatin, external beam radiotherapy, and brachytherapy in patients with stage IB-IVA cervical cancer.

II. Determine the feasibility of this regimen, in terms of chronic and acute toxic effects, in these patients.

SECONDARY OBJECTIVES:

I. Determine the distribution of progression-free survival and overall survival of patients treated with this regimen at 1 year after study entry.

II. Determine the site of recurrence (locoregional vs distant) in patients treated with this regimen up to 1 year after study entry.

III. Correlate response or progression-free survival with epidermal growth factor receptor expression in tumor samples from patients treated with this regimen at 1 year after study entry.

IV. Correlate response or progression-free survival with grade of cetuximab-induced rash in patients treated with this regimen at 1 year after study entry.

OUTLINE: This is a multicenter, dose-escalation study of cetuximab. Patients are stratified according to nodal status (positive para-aortic and/or pelvic lymph nodes vs negative para-aortic and pelvic lymph nodes).

Patients receive cetuximab IV over 1-2 hours and cisplatin IV on days 1, 8, 15, 22, 29, and 36 (weeks 1-6). Patients also undergo external beam radiotherapy to the para-aortic and pelvic lymph nodes OR whole pelvis once daily on days 1-5, 8-12, 15-19, 22-26, and 29-33 (weeks 1-5). Patients then receive either 1 or 2 applications of low-dose rate brachytherapy in weeks 6-8 OR 5 applications of high-dose rate (HDR)* brachytherapy once weekly in weeks 4-8. Treatment continues in the absence of disease progression or unacceptable toxicity.

NOTE: *No external beam radiotherapy is administered on the day of HDR brachytherapy. If the majority of external beam radiotherapy has been administered, HDR brachytherapy may be administered in 2 applications per week (separated by at least 72 hours) in order to complete all treatment within 8 weeks.

Cohorts of 3-6 patients per stratum receive escalating doses of cetuximab until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

After completion of study treatment, patients are followed every 3 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed cervical cancer

  * Clinical stage IB-IVA disease
  * Any cell type allowed
* Positive or negative pelvic and/or para-aortic lymph nodes by radiography
* Unstained sections from primary tumor available
* Performance status - GOG 0-1
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* SGOT ≤ 2.5 times ULN
* Alkaline phosphatase ≤ 2.5 times ULN
* Creatinine normal
* Creatinine clearance > 50 mL/min
* Patients with ureteral obstruction must undergo stent or nephrostomy tube placement prior to study entry
* No renal abnormality (e.g., pelvic kidney or horseshoe kidney) that would require modification of radiation fields
* No significant cardiac disease within the past 6 months, including any of the following:

  * Uncontrolled hypertension
  * Unstable angina
  * Congestive heart failure
  * Uncontrolled arrhythmia
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No sensory or motor neuropathy > grade 1
* No septicemia
* No severe infection
* No circumstance that would preclude study participation or follow-up
* No other invasive malignancy within the past 5 years except nonmelanoma skin cancer
* No uncontrolled seizure disorder
* No active neurologic disease
* No history of active collagen vascular disease
* No prior chimerized or murine monoclonal antibody therapy
* No prior cytotoxic chemotherapy for cervical cancer
* No prior pelvic or abdominal radiotherapy for cervical cancer
* No concurrent intensity modulated radiotherapy
* No prior renal transplantation
* More than 30 days since prior major surgery (excluding diagnostic biopsy)
* No other prior therapy for cervical cancer
* No prior cancer treatment that would preclude study therapy
* No other concurrent investigational agents

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2005-01; Primary Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) or biologically effective dose (BED) of Cetuximab in combination with cisplatin and extended field radiation or whole pelvis radiation, graded using Common Terminology Criteria for Adverse Events version 3.0 (CTCAE v3.0) | 6 weeks
  Evaluation of the regimens will be conducted separately by the type of radiation received (extended field radiation or whole pelvis radiation).
Incidence of toxicities at the MTD, assessed by CTCAE v3.0 | Up to 1 year

SECONDARY OUTCOMES:
Progression-free survival | From study entry until disease progression, death or date of last contact, up to 1 year
Site of recurrence, loco-regional vs distant, assessed by clinical and radiological evaluation | From study entry until disease progression, death or date of last contact, up to 1 year
Frequency of chronic toxicities, assessed by CTCAE v3.0 | From study entry until disease progression, death or date of last contact, up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Moore, Principal Investigator — Gynecologic Oncology Group
Locations (15):
- United States (15):
  - Georgia Regents University Medical Center, Augusta, Georgia
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Johns Hopkins University/Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Lake University Ireland Cancer Center, Mentor, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Women and Infants Hospital, Providence, Rhode Island
  - Parkland Memorial Hospital, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - M D Anderson Cancer Center, Houston, Texas